CLINICAL TRIAL: NCT00958672
Title: Evaluation Des Anomalies Muqueuses Intestinales Par vidéocapsule Endoscopique au Cours de la sclérodermie systémique : Etude Prospective, Multicentrique et Inter-régionale
Brief Title: Small Intestinal Mucosal Abnormalities in Systemic Sclerosis Using Capsule Endoscopy
Acronym: sclero-video
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2008/074/HP
Record Dates: First submitted 2009-07-17; First posted 2009-08-13 (Estimated); Last update posted 2014-06-19 (Estimated); Status verified 2014-06

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Endoscopic capsule — Endoscopic capsule

SUMMARY:
The aim of this prospective study is to determine prevalence and characteristics of small intestinal mucosal abnormalities in 40 patients with systemic sclerosis, using capsule endoscopy. The investigators' findings may improve management of small intestinal involvement in patients with systemic sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Systemic sclerosis based on the ACR diagnostic criteria

Exclusion Criteria:

* Patients with other connective tissue diseases
* Pregnancy
* Absence of contraception in women
* Patients with pace maker
* Patients with intestinal pseudo-obstruction

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 consecutive patients with systemic sclerosis will be included in this prospective study, without prior selection on digestive clinical manifestations
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Prevalence and characteristics of small intestinal mucosal involvement in 40 patients with systemic sclerosis | 1 year

SECONDARY OUTCOMES:
- to assess a correlation between the presence of small intestinal mucosal abnormalities and digestive symptoms | 1 year
to assess a correlation between small intestinal mucosal abnormalities and nutritional status | 1 year
to assess a correlatio between small intestinal mucosal abnormalities and extra-intestinal manifestations of systemic sclerosis | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU-Rouen, Rouen, Rouen, France